CLINICAL TRIAL: NCT05945511
Title: Silent Gallbladder Stone in Kidney Transplantation Recipients: Should it be Treated?
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Woo Hyun Paik, Professor, Seoul National University Hospital
Other Study IDs: 2209-029-1355
Record Dates: First submitted 2023-06-26; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Gallbladder Stones; Kidney Transplantation
MeSH Terms: conditions — Cholecystolithiasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Kidney transplant patients: KT recipients at Seoul national university hospital from January 2005 to July 2022.

SUMMARY:
Treatment and follow-up strategies for silent gallbladder (GB) stones in patients before KT (Kidney transplantation) remain unknown. Therefore, we aimed to assess the risk of gallstone-related biliary complications and post-cholecystectomy complications in KT recipients, to elucidate the role of prophylactic cholecystectomy in this population.

DETAILED DESCRIPTION:
Kidney transplantation (KT) is the best treatment option for patients with end-stage kidney disease (ESKD) although donor deficit remains a main problem. Hence, the survival extension of both KT recipients and their invaluable grafts should be prioritized. A thorough pretransplant evaluation is essential in identifying and managing any risk factors associated with adverse outcomes for both patients and grafts following KT. Candidates typically undergo various types of intra-abdominal imaging before KT surgery to assess the anatomical structures of the renal vasculature and urinary tract, which is crucial for detailed surgery planning and to rule out any pre-existing malignancies or concealed infectious complications. Asymptomatic gallstones may be incidentally discovered during the evaluation, but optimal management and follow-up strategies for these gallstones in KT candidates remain unclear.

Asymptomatic gallstone management in the general population is typically based on the risk of developing relevant symptoms or complications. Previous large cohort studies have revealed that individuals with asymptomatic gallstones have a lifetime risk of approximately 7%-26% of developing serious symptoms or gallstone-related complications such as acute cholecystitis, acute cholangitis, and acute pancreatitis. The aftereffects should not be ignored even if cholecystectomy is performed in patients with asymptomatic gallstones. The incidence of complications after cholecystectomy in the general population is approximately 2.4%-9.4%, and the mortality rate is <1%. Therefore, prophylactic cholecystectomy is not usually recommended in the general population with asymptomatic gallstones.

On the contrary, patients who underwent solid organ transplantation, including KT, had higher rates of both asymptomatic gallstones and postoperative complications after cholecystectomy than the general population. Several studies have revealed that 18%-39% of KT recipients with asymptomatic gallstones develop gallstone-related complications requiring surgery. The postoperative complication rate was approximately 15% and the mortality rate was up to 7% when subsequent cholecystectomy was performed, which indicates an increased morbidity, especially in the case of open surgery. Considering both, the benefit of prophylactic cholecystectomy in KT recipients is difficult to define. Several studies recommend prophylactic cholecystectomy for patients with asymptomatic gallstones who underwent solid organ transplants or those who will require immunosuppressants. Routine cholecystectomy is not typically performed by most transplant centers, despite these recommendations, even when silent gallstones are discovered during the pretransplant evaluation.

Therefore, this retrospective cohort analysis aimed to assess the risk of gallstone-related biliary complications and post-cholecystectomy complications in KT recipients, to elucidate the role of prophylactic cholecystectomy in this population.

ELIGIBILITY:
Inclusion Criteria:

* Kidney transplantation patients

Exclusion Criteria:

1. patients aged <18 years
2. patients followed for <3 months
3. patients without evidence of gallstones on abdominal imaging studies

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Kidney transplantation recipients with gallstones at Seoul national university hospital from January 2005 to July 2022.
Sampling Method: Non-Probability Sample
Enrollment: 2295 (Actual)
Dates: Start 2022-09-07 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-06-01 (Actual)

PRIMARY OUTCOMES:
biliary complications | through study completion, an average of 6 year
  Incidence rate of biliary complication
post-cholecystectomy complications | Within 1month after cholecystectomy
  Incidence rate of post-cholecystectomy complication

SECONDARY OUTCOMES:
Graft failure (GF) | After KT to study completion, an average of 6 year
  Incidence rate of graft failure after kidney transplantation
Death-censored graft failure (DCGF) | After KT to study completion, an average of 6 year
  Incidence rate of Death-censored graft failure after kidney transplantation
All-cause mortality | through study completion, an average of 6 year
  Incidence rate of death

CONTACTS AND LOCATIONS:
Overall Officials: Myeong Hwan Lee, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Lee MH, Jang Y, Kang E, Kim YC, Min S 2nd, Lee SH, Cho IR, Paik WH, Lee H. Silent gallbladder stone in kidney transplantation recipients: should it be treated? A retrospective cohort study. Int J Surg. 2024 Jun 1;110(6):3571-3579. doi: 10.1097/JS9.0000000000001394. PMID 38573083